CLINICAL TRIAL: NCT01213758
Title: Radiation Induced Change of Liver Function Measured by Uptake of the Galactose Analogue FDGal and PET/CT
Brief Title: Changes in Liver Function After Stereotactic Body Radiation Therapy Measured by PET/CT
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: AarhusLiverRadGal
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Hepatocellular Carcinoma; Cholangiocarcinoma; Metastases; Stereotactic Body Radiotherapy
Keywords: liver function; galactose; 18-F-deoxy-galactose; PET/CT; stereotactic body radiation therapy; SBRT
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liver tumors: Patients where stereotactic body radiation therapy is planned for primary or metastatic liver tumors.
  Interventions: Other: Measuring liver function by PET/CT

INTERVENTIONS:
Other: Measuring liver function by PET/CT — Measuring liver function by use of FDGal and PET/CT before, 1 month and 3 months after stereotactic radiotherapy for liver tumors

SUMMARY:
Patients treated with stereotactic radiotherapy for liver tumors undergo PET/CT using the galactose analogue 18-F-deoxy-galactose (FDGal) before and after radiotherapy. This technique provides volumetric mapping of liver function and it allows quantisation of liver function. The method may be used for selection of patients for stereotactic radiotherapy of liver tumors, for determination of radiation induced liver dysfunction and may be included into the treatment planning process of stereotactic radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* liver tumor
* referred for stereotactic radiation therapy
* age > 18 years

Exclusion Criteria:

* Impaired kidney function
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver tumors reffered for stereotactic body radiation therapy
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Uptake of FDGal | Before, 1 month and 3 months after stereotactic radiotherapy
  Volumetric uptake of FDGal can be measured is measured by PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Morten Høyer, MD PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark

REFERENCES:
- See also: The Lundbeck Foundation Centre for Interventional Research in Radiation Oncology — http://www.cirro.dk